CLINICAL TRIAL: NCT04529720
Title: Antibody Persistence at 5 Years After a Single Dose Vaccination of Acellular Pertussis Vaccines Containing Genetically-inactivated Pertussis Toxin
Brief Title: 5-year Follow-up After a Single Dose Acellular Pertussis Vaccination
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: TDA202 5 year follow-up
Record Dates: First submitted 2020-08-20; First posted 2020-08-28 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Pertussis
Keywords: TDA202; acellular pertussis vaccine; antibody persistence at 5 years after vaccination; Pertagen; Boostagen; aP vaccine
MeSH Terms: conditions — Whooping Cough | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Approximately 5 mL whole blood will be processed for serum preparation. Sera obtained will be aliquoted into storage tubes and stored ≤ -30 degree Celsius and shipped to Bionet Human Serology Laboratory. The collected sera will be used for immunogenicity assessment for antibody persistence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acellular pertussis vaccine: Antibody persistence at 5 years after a single dose vaccination of acellular pertussis vaccines (Pertagen;Boostagen;Adacel)
  Interventions: Biological: Biological/Vaccine: Pertagen (aP BioNet); Biological: Biological/Vaccine: Boostagen (TdaP BioNet); Biological: Biological/Vaccine: Adacel

INTERVENTIONS:
Biological: Biological/Vaccine: Pertagen (aP BioNet) — Pertagen (aP BioNet) was produced with a recombinant B pertussis strain that was genetically inactivated by the introduction of mutations (Arg9Lys and Glu129Gly) in the ptx operon of the S1 gene. Each 0.5 mL dose of Pertagen (aP BioNet) contained 5 µg PTgen, 5 µg FHA, and 0.3 mg as aluminium cation.
  The study vaccine will be presented in a single-dose prefilled syringe. Each participant will be received one intramuscular injection in the non-dominant deltoid region.
Biological: Biological/Vaccine: Boostagen (TdaP BioNet) — Boostagen (TdaP BioNet) was produced with a recombinant B pertussis strain that was genetically inactivated by the introduction of mutations (Arg9Lys and Glu129Gly) in the ptx operon of the S1 gene. Each 0.5 mL dose of Boostagen (TdaP BioNet) contained 5 µg PTgen, 5 µg FHA, and 0.3 mg as aluminium cation. TdaP dose additional contained at least 7.5 Lf tetanus toxoid and at least 2.0 Lf diphtheria toxoid.
  The study vaccine will be presented in a single-dose prefilled syringe. Each participant will be received one intramuscular injection in the non-dominant deltoid region.
Biological: Biological/Vaccine: Adacel — Comparator vaccine, Adacel (Sanofi-Pasteur, North York, ON, Canada) was produced chemically inactivated pertussis toxin. Each 0.5 mL dose of Adacel (as comparator vaccine) contained 2.5 µg PTchem, 5 µg FHA, 3 µg pertactin, 5 µg fimbriae types 2 and 3, 5.0 Lf tetanus toxoid, 2.0 Lf diphtheria toxoid and 0.33 mg as aluminium cation.
  The study vaccine will be presented in a single-dose prefilled syringe. Each participant will be received one intramuscular injection in the non-dominant deltoid region.

SUMMARY:
In July 2015-November 2016, a phase II/III randomized, observer-blind,controlled study of two acellular Pertussis vaccines (aP standalone and TdaP combined vaccines) manufactured by BioNet-Asia Co., Ltd. (Bionet) and chemically-detoxified Adacel Tdap vaccine was conducted in Bangkok, Thailand in healthy participants aged 12-17 years (Protocol No. TDA202; http://clinicaltrials.in.th;Study ID:TCTR20150703002). A total of 450 participants were enrolled into the study at 2 study sites (Site No.1:Faculty of Medicine Siriraj Hospital; Site No.2:Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University) with equal number of 225 participants enrolled at each study site. During the study, the participants had been randomized in a 1:1:1 ratio to received intramuscularly a booster dose (0.5 mL) of the study vaccines.

This is further follow-up from TDA202 clinical trial, which was completed on 29 November 2016. Target population for this study is the group of participants who had received one dose of one of the three study vaccines in the TDA202 trial at site VTC and who had completed the study follow-up at 1-year after vaccination (223 subjects).

In this current study, the long-term persistence of pertussis antibodies induced by a booster dose of recombinant acellular Pertussis based vaccines (Pertagen and Boostagen) manufactured by Bionet will be evaluated and compared to the conventional chemically-inactivated Tdap vaccine (Adacel) at 5 years after previously immunized in the TDA202 study.

DETAILED DESCRIPTION:
The study population will included all participants who participated in the TDA202 study at the Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University, Bangkok.

Participants from all 3 vaccine groups (i.e., participants who had received a single dose of one of the 3 study vaccines (Boostagen®, Pertagen®, or Adacel®) and completed 1-year follow-up visit at Day 336±28 days during the TDA202 study will be called in for informed consent process at Visit 1 at approximately 5 years after vaccination (±56 days) based on Vaccination Date in the TDA202 study. Participants aged ≥18 years who have signed the written Informed Consent Form or participants aged less than 18 years who have co-signed the Informed Consent Form with their parent/legal will be screened for general health status (a survey for medical history, immunization history, history of receiving blood, blood component, immunoglobulin, immunosuppressive drugs or systemic corticosteroid and physical examination) and those who fulfill the pre-defined inclusion criteria and do not meet an exclusion criteria will be enrolled into the study.

Once enrolled, a blood sample (approx. 5 mL) will be taken from all participants. After blood collection, this will be considered as study end for all participants. Participants will be offered a licensed influenza vaccine at the end of Visit 1.

Blood samples collected from all participants who have come back for the 5-year follow-up visit (Visit 1) will be processed for serum preparation. Serum samples will be stored at the laboratory at the study site and will be further shipped to BioNet Human Serology Laboratory where immunogenicity testing (ELISA antibodies against Pertussis Toxin (PT), Filamentous hemagglutinin (FHA), Diphtheria Toxin (DT), and Tetanus Toxin (TT) and PT-neutralizing antibody by Chinese Hamster Ovary (CHO) cells assay) will be performed. ELISA testing to detect antibodies against tetanus, diphtheria, and pertussis antigens (PT and FHA) will be performed for all enrolled participants while CHO cells assay to detect PT-neutralizing antibody will be performed only in the same subset of participants who had been selected for PT-neutralizing antibody study in the initial TDA202 study.

The knowledge from this long-term 5-year antibody persistence study will provide supportive data to identify the best alternative acellular pertussis vaccines to conventional chemically-inactivated vaccines for controlling the resurgence of pertussis disease.

Data management and statistical analysis will be performed by Center of Excellence for Biomedical and Public Health Informatics (BIOPHICS), Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for inclusion if ALL of the followings apply at the time of screening:

1. Having participated in the initial TDA202 study, received a single dose of one of the 3 study vaccines, and completed 1-year follow-up visit;
2. Written informed consent is obtained for participants aged ≥18 years, or written informed consent are obtained from participants aged <18 years with their parents/legal guardians, co-signed prior to study entry;
3. Healthy, as established by pertinent medical history and physical examination;
4. Capable of complying with study procedures and willing to provide with a blood sample

Exclusion Criteria:

1. Having received pertussis vaccine since TDA202 study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population for this study is the group of participants who had received one dose of acellular pertussis based vaccine in TDA202 trial at Vaccine Trial Centre (VTC), Faculty of Tropical Medicine, Mahidol University and who had completed the study follow-up at 1 year after vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Anti-PT and Anti-FHA GMTs (IU/ml) changed from baseline at 5 Years After Vaccination in All Evaluable Participants by Vaccine Groups | 5 years after vaccination ± 56 days
  Anti-PT and anti-FHA GMTs (IU/mL) at baseline and 5 years after vaccination as assess by ELISA in all evaluable participants by vaccine groups.
Anti-Tetanus and Anti-Diphtheria GMTs (IU/mL) changed from baseline at 5 Years After Vaccination in All Evaluable Participants in Boostagen (BioNet TdaP BioNet) and Adacel Vaccine Groups | 5 years after vaccination ± 56 days
  Anti-Tetanus and anti-Diphtheria GMTs (IU/mL) between baseline and 5 years after vaccination as assessed by ELISA in all evaluable participants in Boostagen (BioNet TdaP BioNet) and Adacel vaccine groups
Seroconversion Rates as Defined by the Proportion of Participants With Booster Response in Anti-PT and Anti-FHA Antibody Titers at Day 28 and 5 Years After Vaccination Compared to Baseline in All Evaluable Participants by Vaccine Groups | 5 years after vaccination ± 56 days
  Booster response:
  * In initially seronegative subjects (baseline titer < 5 IU/mL), post-vaccination antibody concentrations ≥ 20 IU/mL;
  * In initially seropositive subjects with baseline titer ≥ 5 IU/mL and < 20 IU/mL, an increase of at least 4 times (≥ 4-fold) the baseline titer;
  * In initially seropositive subjects with baseline titer ≥ 20 IU/mL, an increase of at least 2 times (≥ 2-fold) the baseline titer
PT Neutralizing GMTs (IU/mL) changed from baseline at 5 Year After Vaccination as Assessed in a Subset of Evaluable Participants by Vaccine Group | 5 years after vaccination ± 56 days
  PT neutralizing GMTs (IU/mL) between baseline and 5 year after vaccination as assessed by PT neutralizing assay in a subset of evaluable participants by vaccine group
Seroconversion Rates Defined by Proportion of Participants With ≥ 4-fold Changed in PT Neutralizing Antibody Titers at Day 28, Day 336 and 5 Years After Vaccination Compared to Baseline in a Subset of Evaluable Participants | Day 28, Day 336 and 5 years after vaccination ± 56 days
  Seroconversion rates as defined by the proportion of participants with ≥ 4-fold increase in PT neutralizing antibody titers at Day 28, Day 336 and 5 years after vaccination compared to baseline as assessed by PT neutralizing assay in a subset of evaluable participants by vaccine group

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Principal Investigator — VTC, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, 420/6 Ratchawithi Road, Ratchathewi,, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pitisuttithum P, Chokephaibulkit K, Sirivichayakul C, Sricharoenchai S, Dhitavat J, Pitisuthitham A, Phongsamart W, Boonnak K, Lapphra K, Sabmee Y, Wittawatmongkol O, Chauhan M, Wijagkanalan W, Hommalai G, Fortuna L, Chinwangso P, Poredi IK, van den Biggelaar AHJ, Pham HT, Viviani S. Antibody persistence after vaccination of adolescents with monovalent and combined acellular pertussis vaccines containing genetically inactivated pertussis toxin: a phase 2/3 randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2018 Nov;18(11):1260-1268. doi: 10.1016/S1473-3099(18)30375-X. Epub 2018 Sep 25. PMID 30266329